CLINICAL TRIAL: NCT06276283
Title: A Phase II, Single Arm, Multicenter Study to Assess the Safety, Tolerability and Anti-Tumor Efficacy of DZD9008 With Bevacizumab in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Harboring EGFR Mutations (WU-KONG29)
Brief Title: DZD9008 In Combination With Bevacizumab in Locally Advanced or Metastatic NSCLC Patients With EGFR Mutation (WU-KONG29)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2022E0006
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DZD9008 plus Bevacizumab (Experimental): This single-arm study includes two parts (dose escalation [Part A] and dose expansion [Part B]).
  Interventions: Drug: DZD9008 plus Bevacizumab

INTERVENTIONS:
Drug: DZD9008 plus Bevacizumab — DZD9008, 200 mg or 300 mg, once daily plus Bevacizumab 15 mg/kg, once every 3 weeks
  Other Names: Inapplicable

SUMMARY:
This study tests a combination therapy (i.e., DZD9008 plus bevacizumab) in patients with advanced NSCLC harboring EGFR mutations who have progressed on or after standard of care, which aims to understand whether the combination therapy is safe, how well the combination therapy works, and how the body will process DZD9008 when used in combination with bevacizumab.

DETAILED DESCRIPTION:
A phase 2, multicenter study to evaluate the safety, tolerability, and anti-tumor efficacy in patients with locally advanced or metastatic NSCLC harboring EGFR mutations. This study comprises two parts (Part A, dose escalation and Part B, dose expansion). Part A will enroll patients with different EGFR mutations. Only patients with EGFR Exon 20 insertion mutation will be enrolled into Part B.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria for inclusion in the study:

1. Sufficient understanding of nature of the trial and provision of informed consent with hand-written signatures and the date of signature prior to any study-specific procedures, sampling, and analyses.
2. Age ≥ 18 years.
3. Histologically or cytologically confirmed and locally advanced or metastatic non-squamous NSCLC.
4. Written documentation of EGFR mutations from an accredited local laboratory: Part A is not limited to a specific EGFR mutation, and Part B only includes patients with EGFR Exon20ins.
5. ECOG score ≤ 1 without clinically significant disease deterioration within 2 weeks prior to the informed consent process and a life expectancy ≥ 12 weeks.
6. Patients with stable brain metastasis provided no evidence of progression for at least 2 weeks, as ascertained by brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during the screening period, no neurological symptoms, and no requirement of Steroids.
7. Part A includes patients who have progressed after or cannot tolerate the standard of care
8. Part B includes patients with NSCLC who have progressed after or cannot tolerate standard of care. Treatment naïve patients will be enrolled after an adequate evaluation of the safety data by the Safety Review Committee (Note: Patients who have received (neo)adjuvant therapy are allowed to participate in the study, if the (neo)adjuvant therapy is administrated at least 6 months prior to the diagnosis of locally advanced or metastatic NSCLC) .
9. Measurable lesions, according to RECIST 1.1: at least one lesion, not previous irradiated, with the longest diameter ≥ 10 mm at baseline (lymph nodes must have a short axis of ≥ 15 mm), that can be accurately measured at baseline and thereafter with MRI or CT scan.
10. Male patients with a female partner or fertility desire should be willing to use barrier contraception (e.g., condoms) until 6 months after the last dose. Male patients should not donate sperms until 6 months after the last dose. Male patients with fertility desire are suggested to freeze their sperm before entering the study.
11. Female patients should be willing to use adequate contraceptive measures, should not be breastfeeding, and must have a negative pregnancy test (i.e., urine and blood pregnancy human chorionic gonadotropin testing); or female patients meet the following criteria:

    * Post-menopausal defined as age more than 60 and amenorrheic for at least 12 months after all exogenous hormonal treatments.
    * Women under 60 years old would be considered post-menopausal if they have been amenorrheic for at least 12 months with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range.
    * Documentation of irreversible surgical sterilization (e.g., hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation).

Exclusion Criteria:

Patients must not enter the study if any of the following exclusion criteria are met:

1. Treatment with any of the following:

   * Treatment with poziotinib, mobocertinib (TAK788), CLN-081, BDTX-189, aumolertinib, AP-L1898, and other EGFR Exon20ins inhibitors prior to the first dose of study drug (only applicable to Part B).
   * Prior treatment with 1st to 3rd generation EGFR-TKIs (e.g., gefitinib, erlotinib, icotinib, osimertinib, afatinib, dacomitinib, and ametinib) and have had an objective response (i.e., PR and CR) (only applicable to Part B).
   * Prior systemic treatment for locally advanced or metastatic NSCLC (only applicable to treatment naïve patients in Part B)
   * Treatment with EGFR, HER2, or VEGFR antibody within 4 weeks of the first dose of study drug.
   * Chemotherapy or other anti-tumor therapies within 2 weeks of the first dose of study drug.
   * Radiotherapy within 14 days of the first dose of study drug or unresolved radiotherapy-related toxicities. Patients could receive palliative radiotherapy for tumor lesions outside of brain and chest, stereotactic radiosurgery, and stereotactic body radiotherapy.
   * Current treatment within 1-2 weeks of the first dose of study drug with medications or herbal supplements known to be potent inhibitors (1 week) or inducers (2 weeks) of cytochrome P450 (CYP) 3A4.
   * Major surgery, excluding biopsy and diagnostic surgery, within 4 weeks of the dose of study drug, or expected major surgeries during the study period.
   * Treatment with an investigational drug within 5 half-lives of the compound. Patient
2. Spinal cord compression or leptomeningeal metastasis.
3. Concurrent EGFR mutations with approved EGFR-TKIs (e.g., Exon19del, L858R, T790M, G718X, S768I and L861Q; only applicable to Part B).
4. History of malignancy within 2 years of the first dose of study drug (excluding adequately treated Basal cell carcinoma or in situ cervical cancer with a tumor-free period of more than 2 years and a life expectancy of more than 2 years. The inclusion of such patients should be discussed with the study physician from Dizal Pharma).
5. Any unresolved toxicities from prior systemic therapy (e.g., adjuvant chemotherapy and radiotherapy) > CTCAE grade 1 at the time of starting study drug except for alopecia and grade 2 neuropathy related to previous platinum-based therapy.
6. History of stroke and intracranial hemorrhage within 6 months of the first dose of study drug.
7. Any evidence of severe or uncontrolled systematic disease based on the investigator's opinion, including uncontrolled hypertension and active bleeding diatheses (e.g., hemophilia and von Willebrand disease).
8. Any evidence of active infection, including but not limited to hepatitis B, hepatitis C, human immunodeficiency virus (HIV), and COVID-19. The diagnosis of COVID-19 follows the local practice.

   Test Include if Exclude if HIV antibody (-) (+) HCV antibody (-) (+) HBV antibody HbsAg (-) and HbcAb (-) HbsAg (+) and HBV DNA ≥ 1000 IU/mL HbsAg (-), HbcAb (+) and HBV DNA < 1000 IU/mL HbsAg (-), HbcAb (+), and HBV DNA ≥ 1000 IU/mL (-), Negative; (+), Positive.
9. Any of the following cardiac events or abnormalities:

   * Mean resting corrected QT interval (QTcF) > 470 msec.
   * Any clinically significant abnormalities in rhythm, conduction, or morphology detected by resting ECG, e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, and PR interval > 250 msec.
   * Any factors that can lead to QTcF prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, family history of unexplained sudden death under 40 years of age, or any comorbidities known to prolong the QT interval.
   * Any evidence of atrial fibrillation (except for drug-related atrial fibrillation that has been resolved after drug discontinuation).
   * Any evidence of myocadiac infraction, congestive heart failure (New York Heart Association Class II or above), and uncontrolled arrhythmia with medication within 6 months of the first dose of study drug.
10. History of interstitial lung disease (ILD), drug-induced ILD, and immune-related pneumonitis due to cancer immunotherapy.
11. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing the study drug, or previous bowel resection that would preclude adequate absorption of DZD9008.
12. Inadequate bone marrow reserve or organ function:

    * Absolute neutrophil count < 1.5 × 109/L
    * Platelet count < 100 ×109/L
    * Hemoglobin < 9 g/dL
    * Total bilirubin >1.5 × ULN if no liver metastases or >3 × the upper limit of normal (ULN) in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST >2.5 × ULN if no demonstrable liver metastases or >5 × ULN in the presence of liver metastases.
    * Creatinine ≥1.5 × ULN or creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation)
    * The international normalized ratio > 1.5 × ULN and activated partial thromboplastin time (APTT) > 1.5 × ULN
    * Serum lipase) > 1.5 × ULN and serum amylase > 1.5 × ULN
13. Live virus vaccines administrated within 2 weeks of the first dose of study drug.
14. Pregnant women or women who are breastfeeding.
15. Concurrent contraindications to bevacizumab, including but not limited to:

    * Deep vein thrombosis ≥ CTCAE grade 3
    * Uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg)
    * Intracerebral hemorrhage, including hemorrhage caused by metastatic brain tumors.
    * History of severe proteinuria (urine dipstick protein 2+ or 24-hour urine protein > 2g)
    * History of hypertensive crisis and hypertensive encephalopathy
    * History of central nervous system diseases that are not related to the tumor (e.g., convulsions)
    * History of vascular events within 6 months of the first dose of study drug (e.g., aneurysm requiring treatment)
    * History of hemoptysis within 3 months of the first dose of study drug (two spoonfuls of blood each time)
    * History of bleeding disorders or coagulation disorders without treatment of anticoagulants.
    * Tumor invasion of major vessels
    * History of gastrointestinal perforation or fistula within 6 months of the first dose of study drug
16. Severe allergic reaction to DZD9008, bevacizumab, or their excipients.
17. Subjects who are involved in the design, planning, or conduct of the study (applicable to employees of Dizal Pharm and staff at investigational sites).
18. Poor compliance or inability to participate in clinical studies according to the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Part A: 1) Dose Limiting Toxicity (DLT); 2) Treatment-Emergent Adverse Events (TEAEs); TEAEs ≥CTCAE grade 3; and Serious Adverse Events (SAEs). Part B: 1) TEAEs; TEAEs ≥CTCAE grade 3; and SAEs. | The first treatment cycle (each cycle is 21 days) for DLT; From the first dose of study treatment to 28 days after the last dose of study treatment for TEAE; and from ICF signature to 28 days after the last dose of study treatment for SAE.
  To investigate the safety and tolerability of DZD9008 in combination with Bevacizumab in patients with locally advanced NSCLC harboring EGFR mutations. Part A is a dose escalation study to determine the recommended phase 2 combination dose of DZD9008 and Bevacizumab. Part B is a dose expansion study to further investigate the safety and tolerability of the combination therapy at the recommended phase 2 combination dose.

SECONDARY OUTCOMES:
Part A: 1) Tumor response per RECIST 1.1 and 2) Plasma concentration of DZD9008 and its metabolite. Part B:1) Tumor response per RECIST 1.1; 2) Intracranial tumor response per RECISIT 1.1; 3) Plasma concentration of DZD9008 and its metabolite. | From the first dose of study treatment to disease progression, death or study withdrawal, whichever occurs first; and Cycle 1/3/5/7 day 1 (each cycle is 21 days) for plasma concentration of DZD9008 and its metabolite.
  To investigate the anti-tumor efficacy of DZD9008 in combination with Bevacizumab and the pharmacokinetics of DZD9008 and its metabolite DZ0753 when given in combination with Bevacizumab. The efficacy endpoints per RECIST 1.1 include Objective Response Rate (ORR), Duration of Response (DoR),Disease Control Rate (DCR), and Progression Free Survival (PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Lu, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No